CLINICAL TRIAL: NCT00115258
Title: Nutrition Support in Pediatric Stem Cell Transplantation - A Randomized, Controlled Trial
Brief Title: Nutrition Support in Pediatric Stem Cell Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Christopher Duggan, Associate professor of pediatrics, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 86483; 03-11-192
Record Dates: First submitted 2005-06-21; First posted 2005-06-22 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Hematopoietic Stem Cell Transplantation
Keywords: Nutrition, Parenteral; Body Composition; Energy Expenditure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- parenteral nutrition titrated to measured REE (Experimental): parenteral nutrition titrated to measured REE
  Interventions: Other: parenteral nutrition titrated to measured REE
- standard of care (No Intervention)

INTERVENTIONS:
Other: parenteral nutrition titrated to measured REE
  Arms: parenteral nutrition titrated to measured REE

SUMMARY:
The purpose of this study is to determine which method of providing parenteral nutrition (complete intravenous nutrition) will provide the best nutritional and clinical results to children undergoing hematopoietic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* First myeloablative allogeneic SCT using either TBI (1400 cGy) or busulfan in addition to other chemotherapeutic agents
* GVHD prophylaxis with a calcineurin-inhibitor and methotrexate +/- corticosteroids
* Matched, related or 6/6 HLA-matched unrelated SCT donor
* Age 6 years and older

Exclusion Criteria:

* Age less than 6 years, or otherwise unable to comply with study procedures
* Underweight (body mass index (BMI) z-score <2 for age and sex) at baseline
* Overweight (BMI z-score >2 for age and sex) at baseline
* Unable or unwilling to return for day + 100 studies
* Previous stem cell transplant
* Unmatched SCT donor
* Current treatment for hypo- or hyperthyroidism
* Current insulin dependent diabetes
* Current use of parenteral nutrition
* Allergy to egg or soy products
* Other contraindication to parenteral nutrition at baseline

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2004-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Changes in % body fat at baseline, day +30, and day +100. | day 30

SECONDARY OUTCOMES:
Body composition measured by DXA, BIA, and 4-site skinfolds. | baseline, day 30, and day 100
Changes in body composition from baseline to day +100. | day 100
Insulin resistance, defined by HOMA, at each time point. | baseline, day 30, and day 100
Measured resting energy expenditure (REE) at each time point. | baseline, day 30, and day 100
Changes in percent predicted REE between the two groups. | baseline, day 30, and day 100
Correlation between body composition and measured REE. | baseline, day 30, and day 100
Resumption of oral intake. | day 30

CONTACTS AND LOCATIONS:
Overall Officials: Christopher P. Duggan, M.D., M.P.H., Principal Investigator — Boston Children's Hospital

REFERENCES:
- [Background] Duggan C, Bechard L, Donovan K, Vangel M, O'Leary A, Holmes C, Lehmann L, Guinan E. Changes in resting energy expenditure among children undergoing allogeneic stem cell transplantation. Am J Clin Nutr. 2003 Jul;78(1):104-9. doi: 10.1093/ajcn/78.1.104. PMID 12816778
- [Background] Bechard LJ, Feldman HA, Gordon C, Gura K, Sonis A, Leung K, Venick R, Guinan EC, Duggan C. A multi-center, randomized, controlled trial of parenteral nutrition titrated to resting energy expenditure in children undergoing hematopoietic stem cell transplantation ("PNTREE"): rationale and design. Contemp Clin Trials. 2010 Mar;31(2):157-64. doi: 10.1016/j.cct.2009.12.002. Epub 2010 Jan 3. PMID 20004739
- [Result] Sharma TS, Bechard LJ, Feldman HA, Venick R, Gura K, Gordon CM, Sonis A, Guinan EC, Duggan C. Effect of titrated parenteral nutrition on body composition after allogeneic hematopoietic stem cell transplantation in children: a double-blind, randomized, multicenter trial. Am J Clin Nutr. 2012 Feb;95(2):342-51. doi: 10.3945/ajcn.111.026005. Epub 2011 Dec 28. PMID 22205317